CLINICAL TRIAL: NCT05486260
Title: Effect of Regular Consumption of Dried Miracle Berry (DMB) on Taste Perception and Nutritional Status in Malnourished Cancer Patients: A Triple-Blind, Randomized, Placebo-Controlled Clinical Trial. CLINMIR Pilot Protocol
Brief Title: Effect of Dried Miracle Berry on the Olfactory-gustative Perception in Malnourished Cancer Patients
Acronym: CLINMIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other); Medicinal Gardens S.L (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HULP 6164
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-05

CONDITIONS: Cancer; Dysgeusia; Hypogeusia; Ageusia; Chemotherapy Effect; Malnutrition
MeSH Terms: conditions — Neoplasms; Dysgeusia; Ageusia; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Pills with 300 mg of DMB equivalent to 5,5 mg of the miraculin glycoprotein
  Interventions: Dietary Supplement: DMB highest dose
- Group B (Experimental): Pills with 150 mg of DMB equivalent to 2,8 mg of miraculin glycoprotein + 150g of freeze-dried strawberry
  Interventions: Dietary Supplement: DMB lowest dose
- Group C (Placebo Comparator): Pills with 300 mg of strawberry lyophilisate
  Interventions: Dietary Supplement: Strawberry lyophilisate

INTERVENTIONS:
Dietary Supplement: DMB lowest dose — Intake of 150 mg of DMB
  Other Names: Experimental 1
  Arms: Group B
Dietary Supplement: DMB highest dose — Intake of 300 mg of DMB
  Other Names: Experimental 2
  Arms: Group A
Dietary Supplement: Strawberry lyophilisate — Intake of 300 mg of strawberry lyophilisate
  Other Names: Placebo comparator
  Arms: Group C

SUMMARY:
Cancer is one of the main causes of death globally, being in many countries the first cause of mortality. One of the main side effects of chemotherapy and/or radiotherapy treatment in cancer patients is the alteration of taste and smell, internationally known as these anomalies Taste Smell Alterations (TSA). These alterations are the result of an altered cellular structure, the presence of TSA is associated with reduced quality of life and poor nutrition, due to dietary changes made by these patients.

Synsepalum dulcidicum (dried miracle berry, DMB) is a plant belonging to the Sapotaceae family, made up of around 800 species grouped into around 40 genera. It is an indigenous species to the forest regions of West Africa. Nuts of this specie have been approved as a novel food in accordance with Regulation (EU) 2015/2238 and at the request of the European Commission through the European Food Safety Authority (EFSA) Panel on Nutrition, Novel Foods and Food Allergens. The characteristic component of DMB is miraculin. Miraculin is a glycoprotein whose consumption causes acidic and sour foods, and to a lesser extent bitter, to be perceived as having a sweet taste. In this sense, it is possible that the consumption of DMB before each meal can improve sensory perception after treatment with chemotherapy or radiotherapy.

DETAILED DESCRIPTION:
Randomized, parallel, triple-blind, controlled clinical trial to evaluate the effect of habitual consumption of DMB on the olfactory-gustative perception in cancer patients with malnutrition.

30 volunteers will be recruited at the La Paz University Hospital of Madrid. Participants should meet the next inclusion criteria: men and women over 18, a weight loss >=5 %, malnutrition, taste alterations, cancer patients treated with neoadjuvant chemotherapy prior to surgery, chemotherapy or chemo-radiotherapy who are not candidates for surgery, with less than or equal to one third of chemotherapy and/or radiotherapy treatment initially scheduled, a life expectancy greater than 3 months, oral intake of food and drinks, adequate cultural level and understanding of the clinical study.

Participants will be randomized in 3 arms:

1. Group A (150mg de DMB equivalent to 2, 8 mg of miraculin glycoprotein + 150g of freeze-dried strawberry).
2. Group B (300 mg of DMB equivalent to 5, 5 mg of the miraculin glycoprotein).
3. Group C (300 mg of strawberry lyophilisate).

   Follow up will include 6 individualized visits, to perform the following tests at each visits:

   Selection visit

   • Nutritional assessment

   • Electrogustometry

   • Olfactory-gustative test (test strips)
   * Taste and smell survey.

     1º visit:
   * Measurement of blood pressure and heart rate
   * Morphofunctional assessment:

     o Anthropometry measures (weight, % weight loss, height, BMI, ICA)

     o Bioelectrical impedance (BIA): musculoskeletal mass index (MMI), phase angle (FA), extracellular water (EW), intracellular water (IW) and total water (TBW), fat mass (FM), muscle mass (MM), total cell mass, representation phase angle vector (BIVA)

     o Dynamometry

     o Nutritional ultrasound

     o Functionality test (Up and Go Test)
   * Olfactory-gustative test (Sniffin'Stick Smell Test)
   * Saliva volume.
   * Analytic:

     o Biochemistry (albumin, prealbumin, retinol-binding protein (RBP), glucose, lipid profile (Total Cholesterol (TC), triglycerides (TG), HDL, LDL), safety parameters (transaminases, urate, creatinine), fat-soluble vitamins (A, D, E), B12, folate, iron metabolism, Zn, Se. Hemogram, lymphocytes, coagulation, hsCRP)

     o Stool microbiota and metagenome

     o Saliva microbiota and metagenome

     o Plasma metabolomes

     o Quantitative profile of fatty acids in erythrocytes (enzymatic activity of catalase (CAT), superoxide dismutase (SOD), glutathione-reductase (GR) and glutathione peroxidase (GPOX))

     o Plasma cytokine profile (Interleukin (IL) 1β, 4, 6, 8, 10 tumor necrosis factor (TNFα), interferon γ (IFNγ), sIL6R, sTNFR)

     o Metabolites in urine

     o System status of antioxidant status (hydroxyguanosine and F2-Isoprostanes)

     2º visit:
   * Anthropometric measures
   * Electrogustometry
   * Olfactory-gustative test
   * Saliva volume
   * Taste and smell survey
   * Product efficacy satisfaction questionnaire (post-QTx)

     3º and 4º visit:
   * Morphofunctional assessment:
   * Measurement of blood pressure and heart rate,
   * Electrogustometry
   * Olfactory-gustative test
   * Saliva volume
   * Taste and smell survey
   * Product efficacy satisfaction questionnaire (pre-QTx)
   * Analytic:

     o Biochemistry

     o Stool microbiota and metagenome (v3)

     o Saliva microbiota and metagenome

     o Plasma metabolomes

     o Quantitative profile of fatty acids in erythrocytes

     o Plasma cytokine profile

     o Metabolites in urine

     o System status of antioxidant status

     5º visit:
   * Morphofunctional assessment:
   * Measurement of blood pressure and heart rate,
   * Electrogustometry
   * Olfactory-gustative test
   * Saliva volume
   * Taste and smell survey
   * Product efficacy satisfaction questionnaire (pre-QTx)
   * Analytic:

     o Biochemistry

     o Stool microbiota and metagenome (v3)
     * Saliva microbiota and metagenome
     * Plasma metabolomes
     * Quantitative profile of fatty acids in erythrocytes
     * Plasma cytokine profile
     * Metabolites in urine
     * System status of antioxidant status

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18
* Patients with a weight loss >=5 %
* Patient with malnutrition assessed by Global Leadership Initiative on Malnutrition (GLIM) Criteria
* Patients with taste alterations measured by electrogustometry
* Cancer patients treated with neoadjuvant chemotherapy prior to surgery, chemotherapy or chemo-radiotherapy who are not candidates for surgery.
* Patients with less than or equal to one third of chemotherapy and/or radiotherapy treatment initially scheduled.
* Patients with a life expectancy greater than 3 months.
* Patient with oral intake of food and drinks.
* Adequate cultural level and understanding of the clinical study.
* Agree to voluntarily participate in the study and give their signed written informed consent.

Exclusion Criteria:

* Patients who are participating in other clinical trials.
* Patients with a weight loss < 5%
* Patients with a parenteral o enteral nutrition
* Patients diagnosed with poorly controlled Diabetes Mellitus (HbA1 c>8%)
* Patients with uncontrolled high blood pressure.
* Patients with uncontrolled hyper/hypothyroidism.
* Patients with severe digestive toxicity due to treatment with chemo-radiotherapy
* Patients with a life expectancy of less than 3 months.
* Patients diagnosed with severe kidney or liver disease (chronic kidney failure, nephrotic syndrome, cirrhosis).
* Patients with severe dementia, brain metastases, eating behavior disorders, history of serious neurological or psychiatric pathology that may interfere with treatment.
* Patients suffering from alcoholism or substance abuse that may interfere with adherence to treatment.
* Patients with serious gastrointestinal diseases.
* Patients who reject the consumption of DMB.
* Pregnant or lactating women.
* Assessment that, in the clinician's opinion, prevents the patient from participating (severity, etc.)

Withdrawal Criteria:

- Intolerance to the consumption of DMB or Placebo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Electrogustometry | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  In this test, perception thresholds are obtained by electrical stimulation (current in microamperes), administered in different tongue regions through small disc-shaped monopolar electrodes.Three areas of the tongue (fenced papillae, tongue apex, and soft palate) are stimulated on both the right and left sides in ascending order two at a time from -6 dB (4 mA) to 34 dB (400 mA). ) in intervals of 0.5, 1, 1.5 and 2 s. If the stimulus is not detected, a single stimulus will be performed at 36 dB and another at -6 dB, to which the subject must answer whether or not they have been able to detect the stimulus.
Sniffing Stick Smell Test | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Sniffing Sticks are markers filled with an odorous fragrance that when removed from the stick releases the smell.To perform all tests, the open pen is held approximately 2 cm in front of the nostrils and the subject is verbally warned to smell it (for example, by saying the number on the pen). The pens are labeled with red numbers from 1 to 16.
  If the patient hits less than 8 smells, it is considered that they have altered taste and smell
Strips' Test | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Test for the identification of taste deficiencies validated. This test uses spoon-shaped flavor-impregnated filter papers that allow them to be selectively applied to specific areas of the tongue. In this test, 4 flavors (sweet, salty, bitter and acid) are evaluated at 4 different concentrations. The sweet taste will be represented by sucrose (0.4, 0.02, 0.1, 0.05 g/mL), the acid by citric acid (0.3, 0.16, 0.09, 0.05 g/mL), the balance by sodium chloride (0.25, 0.1, 0.004, 0.016 g/dL) and quinine bitter (0.006, 0.0024, 0.0009, 0.0004 g/dL). A 1 is marked if the flavor is detected and a 0 if it is not detected. To obtain the global impression of the taste function, a taste score is performed based on the minimum concentration detected and the flavor used.
Taste and Smell Survey | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  This test is used to explore the prevalence, characteristics, and severity of taste and smell changes in a disease. It is made up of 12 items, 7 of them related to taste and 5 related to smell. For each of the questions, 1 point will be assigned for each question answered negatively. An additional point will be awarded for mild/moderate or rarely/sometimes and 2 points for severe/disabling or often/always. Changes in taste were scored from 0 (no change) to 10 (multiple severe changes) and changes in smell from 0 (no change) to 5 (multiple severe changes).

SECONDARY OUTCOMES:
Weight (kg) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  It is measured using a digital scale for clinical use (capacity 0-150 kg), with the person positioned with their back to the viewer, without shoes, wearing a minimum of warm clothing (pants and t-shirt), heels together, looking forward and posture straight body.
Waist circumference (cm) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The subject assumes a position with arms crossed at the chest. The perimeter is taken at the narrowest level, between the lower costal margin (10th rib) and the iliac crest. The anthropometrist stands in front of the subject, who has his arms slightly abducted, to allow the waist to run around the abdomen. Values greater than 80 centimeters (women) and 94 centimeters (men) are considered a risk for cardiovascular diseases.
Body Mass Index (kg/m2) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  It is the relationship between the individual's body weight (kg) and height (m) squared: Weight/Height2. Values greater than 24,9 kg/m2 are considered as overweight
Manual dynamometry | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  It is assessed by using a dynamometer. The maximum manual pressure force exerted on both hands is assessed three times alternately and the average of these results is obtained.
Muscle ultrasound | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The measurement of muscle thickness loss is performed using a linear transducer with high-frequency sound waves (1-10 MHz).Gray-scale ultrasonography is used with a linear transducer with a coefficient of variation of 1.3%. This measurement includes the vastus medialis and rectus femoris muscles.
Up and go test | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Balance evaluation scale. The patient should sit in the chair with their back supported and their arms resting on the armrests. Ask the person to get up from a standard chair and walk a distance of 3 meters. Have the person turn around, walk back to the chair, and sit back down. Timing begins when the person begins to get up from the chair and ends when they return to the chair and sit down.
Saliva volume (mL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The salivary flow rate is determined. To do this, the amount of saliva collected is weighed in a special plastic container in which volumes are indicated every 0.5 mL up to 5 mL.
Albumin serum concentration (g/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in serum albumin concentration. The normal range is 3.4 to 5.4 g/dL (34 to 54 g/L)
Prealbumin serum concentration (mg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in serum prealbumin concentration. Normal results in adults range between 15 and 36 milligrams per deciliter (mg/dL) or 150 and 360 milligrams per liter (mg/L)
Glucose serum concentration (mg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in fasting serum glucose concentration. The levels are between 74 and 100 mg/dL.
Total Cholesterol serum concentration (mg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in total cholesterol concentration. A concentration less than 200 mg/dL is recommended, with a normal upper limit between 200 and 239 mg/dL. Measurements above 240 mg/dL indicate excessive consumption through diet or familial hypercholesterolemia
Triglycerides serum concentration (mg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in triglyceride concentration. Normal values are less than 150 mg/dL; the upper limit is between 150 and 199 mg/dL. However, values between 200 and 499 mg/dl are considered high or very high (above 500 mg/dl).
LDL-cholesterol serum concentration (mg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in LDL-cholesterol concentration. Optimal levels are less than 100 mg/dL, although concentrations between 100 and 129 mg/dL are considered almost optimal. The upper limit of normal is between 130 and 159. Values between 160 and 189 mg/dL are considered high, and those above 190 mg/dL as very high.
HDL-cholesterol serum concentration (mg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in HDL-cholesterol concentration. Values above 60 mg/dL are considered a protective factor against cardiovascular diseases. Concentrations between 40 and 59 mg/dL are correct, while values below 40 mg/dL are one of the main risk factors for cardiovascular disease.
RCP-us serum concentration (mg/L) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in hs-CPR concentration. It has been shown that hs-CPR provides information on each of the levels of cardiovascular risk according to the Framingham scale; CPR-us levels less than 1 mg/L, between 1 and 3 mg/L, and greater than 3 mg/L, correspond to low, medium, and high cardiovascular risk, respectively.
Vitamin A serum concentration (μg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in Vitamin A concentration. Normal values range from 20 to 60 micrograms per deciliter (mcg/dl) or 0.69 to 2.09 micromoles per liter (micromol/l).
Vitamin D serum concentration (ng/mL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the concentration of Vitamin D. Normal values are 75-100 nmol/L (30-40 ng/ml). Vitamin D deficiency occurs if serum levels of hydroxyvitamin D are less than 50 nmol/L (20 ng/ml), an insufficiency of 50-75 nmol/L (20-30 ng/ml).
Vitamin E serum concentration (alfa-tocopherol, μg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the concentration of Vitamin E as alpha-tocopherol. Normal adult concentrations of alpha tocopherol in plasma or serum are within the range of 500-1600 μg/dL, in preschool children concentration ranges have been proposed to be 300-900 μg/dL.
Vitamin B12 serum concentration (pg/mL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the concentration of Vitamin B12. Normal values are 200 to 900 pg/ml (picograms per milliliter).
Folic acid serum concentration (ng/mL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in serum folic acid concentration. The normal range is 2.7 to 17.0 nanograms per milliliter (ng/mL), or 6.12 to 38.52 nanomoles per liter (nmol/L).
Iron serum concentration (μg/dL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in serum iron concentration. Normal values range from 60 to 170 micrograms per deciliter (μg/dL), or 10.74 to 30.43 micromoles per liter (μmol/L).
Zinc serum concentration (μg/mL) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in serum zinc concentration. The most accepted ranges in clinical trials are between 0.75 and 1.30 μg/mL.
Selenium serum concentration (μg/L) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in serum selenium concentration. Levels between 60 and 100 µg/L are considered normal. Values less than 59.24 µg/L (<0.75 mumol/L) are considered low.
Plasma cytokine concentration | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in plasma cytokine concentrations. They will be determined using the Luminex®200™ multianalyte profile analyzer and the HCYTO-60K-PMX Milliplex Map Kit immunoassay kit. Mean Fluorescent Intensity data will be fitted using the spline or logistic curve-fitting method. 5 parameters to calculate cytokines/chemokines.
Saliva microbiota | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Complete amplicons corresponding to the amplification of the bacterial 16S rRNAr gene will be analyzed.
Saliva metagenomics | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  DNA amplification will be carried out by PCR of the 16S rRNA gene using bacteria-specific primers and adapter-binding barcoding (library preparation). Bacterial DNA sequencing will be analyzed following sequencing standards (IHMS SOPs 08, 09 and 10 V1).
Faeces microbiota | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  DNA amplification will be carried out by PCR of the 16S rRNA gene using bacteria-specific primers and adapter-binding barcoding (library preparation). Bacterial DNA sequencing will be analyzed following sequencing standards (IHMS SOPs 08, 09 and 10 V1).
Faeces metagenomics | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The amplified (sequencing) bacterial DNA will be analyzed following the sequencing standards (IHMS SOPs 08, 09 and 10 V1) and the sequencing data will be further analyzed against the data analysis standards (IHMS SOPs 11).
Plasma metabolomics | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  For the metabolomic analysis, a multiple strategy (EureCat's GlobalMet) will be used for the separation and evaluation of both water-soluble and fat-soluble plasma metabolites (lipidomics) based on semi-directed analysis using GLC-MS (plasma metabolome analysis, non-directed analysis using UPLC-MS and directed analysis by UPLC-MS.
Quantitative profile of fatty acids in erythrocytes | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in fatty acid methyl esters are identified and quantified by comparison of retention times with those of previously used authentic standards and confirmed by mass spectrometry (MS).
Concentration of 8-iso-PGF2α in urine | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The concentration of 8-iso-PGF2α in urine is determined by a highly specific and validated enzyme-linked immunosorbent assay (ELISA). The cross-reactivity of 8-iso-PGF2α antibody with 15-keto-13, 14-dihydro-8-iso-PGF2α, 8-iso-PGF2β, PGF2α, 15-keto-PGF2α, 15-keto-13, 14-dihydro -PGF2α, TXB2, 11β-PGF2α, 9β-PGF2α and 8-iso-PGF3α is 1.7, 9.8, 1.1, 0.01, 0.01, 0.1, 0.03, 1.8 and 0.6%, respectively. The limit of detection of the assay is 23 pmol/L
Concentration of 8-hydroxy-2'-deoxyguanosine in urine | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The concentration of 8-OHdG in urine is determined by an enzyme-linked immunosorbent assay (ELISA) kit. The absorbance at 450 nm is determined with a microplate reader. The determination range is 0.125-10 ng/ml. The 8-OHdG concentration is adjusted for urinary creatinine levels and is expressed as ng 8-OHdG/mg creatinine.
Total antioxidant capacity (TAC) of plasma | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in TAC are evaluated using a spectrophotometric antioxidant assay kit.
Determination of oxidized and reduced glutathione in erythrocytes | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in oxidized and reduced glutathione in erythrocytes determined using a colorimetric technique. GSH concentration can be determined from an end point reading of the color developed at 405nm or by measuring the rate of color development at 405nm.
Enzyme activity of the antioxidant defense system in erythrocytes | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the hemoglobin (Hb) concentration of the samples are determined spectrophotometrically using a colorimetric method. The reading is done at 540 nm and a standard curve is used to calculate the concentration of Hb in the samples (0.08-08 mg/ml).
CAT catalase activity (EC 1.11.1.6) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes are determined by the H2O2 activated fluorescence method. In the ultraviolet (UV) range, H2O2 is characterized by a continuous increase in absorption parallel to a decrease in wavelength (λ). The decomposition of H2O2 is determined by the decrease in absorbance at 240 nm. The difference in absorbance with respect to a blank per unit of time is the measure of CAT activity, which is expressed as nmol/g Hb
SOD superoxide dismutase activity (EC 1.5.1.1) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The changes are determined by the use of xanthine and xanthine oxidase to generate O2 · ̄ radicals, which, in turn, oxidize cytochrome c, generating color that can be measured at 450 nm. Results are expressed as U/mg Hb.
Glutathione Reductase Activity GR (EC 1.6.4.2) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The changes are determined by measuring the rate of oxidation of NADPH in the presence of GSSG. The decrease in absorbance at 340 nm is determined. One unit of enzyme activity is defined as the amount of GR that catalyzes the transformation of 1 μmol of NADPH per min. Results are expressed as U/g Hb.
GPOX glutathione peroxidase activity (EC 1.11.1.9) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes are determined by the coupled reaction of the enzyme with tert-butyl hydroperoxide (t-BOOH) as substrate. The absorbance at 340 nm is measured. In the presence of GR and NADPH, GSSG is immediately converted to GSH along with the oxidation of NADPH to NADP+. One unit of enzyme activity is defined as the amount of GPOX that catalyzes the transformation of 1 μmol of NADPH per min. The results are expressed in U/g Hb.
72 hour food record questionnaire | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Questionnaire to find out the nutritional and dietary habits of each participant. The volunteer will write down all the food and drinks ingested over 3 days (72 hours), considering two school days and one holiday. The answers will allow calculating the total amount of food consumed and calories ingested. In addition, the data will be evaluated quantitatively and qualitatively, classifying the diet in terms of diversity and balance following the recommendations of the Spanish Society of Community Nutrition (SENC 2016).
Food Frequency Consumption Questionnaire (PREDIMED) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Questionnaire to determine the frequency of food consumption. This is evaluated through 9 categories: milk and dairy products; eggs, meat and fish; greens and vegetables; fruits; legumes, cereals and potatoes; oils and fats; pastries and pastries; sauces, fried foods, snacks, sugars and salt; beverages. The subject will record the number of food servings consumed in the last 3 months either per month, per week or per day.
International Physical Activity Questionnaire (IPAQ) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  The questionnaire is divided into 4 categories of questions depending on the type of activity for which information is requested (vigorous, moderate, walking, sedentary). The quantitative results allow calculating the TOTAL Energy Metabolism Rate (MET) x minute/week for each subject. Qualitative results categorize the volunteers' physical activity into low activity (1), moderate activity (2), or vigorous activity (3).
Quality of Life Questionnaire (EORTIC QLQ-C30) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Questionnaire composed of 30 questions or items that assess the quality of life in relation to physical, emotional, social aspects and the level of functionality in cancer patients. For the calculation of this questionnaire, values between 1 and 4 points are assigned, being 1: absolute, 2: little, 3: quite a lot and 4: a lot. The last two items, 29 and 30, are given a score from 1 to 7, with 1: terrible and 7: excellent.
  All scores obtained are standardized. A score of 0 to 100 points is obtained that determines the impact of the disease on the patient for each of the scales. High values in the global health and function scales indicate a better quality of life, while in the symptoms scale it would indicate a decrease in the quality of life since it indicates the presence of cancer-associated symptoms.
Product Efficacy Satisfaction Questionnaire | Before chemotherapy, After therapy (3-4 days), Follow up (3 months after chemotherapy)
  Questionnaire prepared to determine the efficacy of the product by the patient. The survey is based on 6 questions that assess the quality and efficacy of the product by the patient from 0 to 100 points.
Fat mass (%) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the percentage (%) of Fat Mass via bioelectrical impedance
Muscle mass (%) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the percentage (%) of Muscle Mass via bioelectrical impedance
Extracellular water(%) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the percentage (%) of Extracellular Water via bioelectrical impedance
Intracellular water (%) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the percentage (%) of Intracellular Water via bioelectrical impedance
Total Body Water (%) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the percentage (%) of Total Body Water via bioelectrical impedance
Phase angle (º) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the phase angle (grades) via bioelectrical impedance
Body Cell Mass (%) | Before chemotherapy, After therapy (3-4 days), Follow up (1 month, 2 months and 3 months after chemotherapy)
  Changes in the percentage (%) of Body Cell Mass via bioelectrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Samara Palma-Milla, MD, PhD, Principal Investigator — Instituto de Investigación Hospital Universitario La Paz
Locations (1):
- Bricia LOPEZ PLAZA, Madrid, Spain

REFERENCES:
- [Result] Lopez-Plaza B, Gil A, Menendez-Rey A, Bensadon-Naeder L, Hummel T, Feliu-Batlle J, Palma-Milla S. Effect of Regular Consumption of a Miraculin-Based Food Supplement on Taste Perception and Nutritional Status in Malnourished Cancer Patients: A Triple-Blind, Randomized, Placebo-Controlled Clinical Trial-CLINMIR Pilot Protocol. Nutrients. 2023 Nov 1;15(21):4639. doi: 10.3390/nu15214639. PMID 37960292
- [Derived] Alvarez-Mercado AI, Lopez-Plaza B, Plaza-Diaz J, Arcos-Castellanos L, Ruiz-Ojeda FJ, Brandimonte-Hernandez M, Feliu-Batlle J, Hummel T, Palma-Milla S, Gil A. Miraculin Can Contribute to a Reduction in Inflammatory Biomarkers and Cachexia in Malnourished Patients with Cancer and Taste Disorders. Pharmaceuticals (Basel). 2025 Apr 25;18(5):622. doi: 10.3390/ph18050622. PMID 40430444
- [Derived] Lopez-Plaza B, Alvarez-Mercado AI, Arcos-Castellanos L, Plaza-Diaz J, Ruiz-Ojeda FJ, Brandimonte-Hernandez M, Feliu-Batlle J, Hummel T, Gil A, Palma-Milla S. Efficacy and Safety of Habitual Consumption of a Food Supplement Containing Miraculin in Malnourished Cancer Patients: The CLINMIR Pilot Study. Nutrients. 2024 Jun 17;16(12):1905. doi: 10.3390/nu16121905. PMID 38931260